CLINICAL TRIAL: NCT04947852
Title: Efficacy of NIV Masks in COPD Patients With Chronic Respiratory Failure: A Randomized Controlled Cross Over Pilot
Brief Title: Efficacy of NIV Masks in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CIA293
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigation Mask (Experimental): Bi Level CPAP Mask
  Interventions: Device: Investigation Mask; Device: Comparator Mask
- Comparator Mask (Active Comparator): Bi Level CPAP Mask
  Interventions: Device: Investigation Mask; Device: Comparator Mask

INTERVENTIONS:
Device: Investigation Mask — Oronasal bilevel continuous positive airway pressure mask fitted by the investigational staff
Device: Comparator Mask — Oronasal bilevel continuous positive airway pressure mask fitted by the investigational staff

SUMMARY:
A randomized controlled pilot study to compare the efficacy and tolerability of a two different NIV masks on carbon dioxide in participants with stable chronic obstructive pulmonary disease (COPD) with chronic type II respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* A doctor's diagnosis of COPD
* PtCO2 ≥45mmHg on transcutaneous monitor at baseline measure
* Oxygen saturation measured by pulse oximetry (SpO2) ≥85%
* Fits the study mask
* Can tolerate the therapy

Exclusion Criteria:

* FEV1/FVC ≥70%
* Body mass index >35
* Hypercapnia considered to be primarily due to Obesity Hypoventilation syndrome and/or Obstructive Sleep Apnea
* Any condition which makes NIV contra-indicated as per BTS guidelines based on clinical judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Transcutaneous Carbon Dioxide | 60 minutes
  mmHg

SECONDARY OUTCOMES:
Oxygen Saturation | 60 minutes
  Percentage
Minute Ventilation | 60 minutes
  Litres
Heart Rate | 60 minutes
  Beats per minute
Respiratory Rate | 60 minutes
  Breaths per minute
Borg Dyspnoea Score | 60 Minutes
  1-6 Ranking, with 1 being best and 6 being worst

CONTACTS AND LOCATIONS:
Overall Officials: Alex Semprini, Principal Investigator — Medical Research Institute of New Zealand
Locations (1):
- Medical Research Institute New Zealand, Wellington, New Zealand

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.